CLINICAL TRIAL: NCT02336126
Title: Biopsychological Intervention in Chronic Fatigue Syndrome - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIOPSYCH
Record Dates: First submitted 2014-08-22; First posted 2015-01-12 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2015-01

CONDITIONS: Adolescent Chronic Fatigue Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biopsychological intervention (Experimental)
  Interventions: Behavioral: Biopsychological intervention

INTERVENTIONS:
Behavioral: Biopsychological intervention

SUMMARY:
This is a pilot study of a biopsychological intervention program for adolescent chronic fatigue syndrome. The program is related to cognitive behavioral therapy, which has been proven beneficial in this disorders, but includes other mental techniques, such as emotional control and metacognitive elaboration.

The aim of this pilot study is to explore a) patients' experiences and b) possible positive effects on symptoms. We hypothesise that the intervention will be regarded feasible by the patients, and that fatigue score will improve during the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic fatigue syndrome
* Significant school absenteeism
* Above 12 years of age and below 18 years of age

Exclusion Criteria:

* Other diseases or life events that might explain chronic fatigue
* Bed-ridden

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Chalder fatigue score | Up to 3 months after inclusion

SECONDARY OUTCOMES:
Patients' experiences (semistructured interview) | Up to 3 months after inclusion
  Qualitative data, further analysed by thematic structural analysis
Quality of Life (PedsQL) | Up to 3 months after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Akershus university hospital, Lørenskog, Akershus, Norway